CLINICAL TRIAL: NCT06301867
Title: Preventing Failed Extubations Cohort Study
Brief Title: Preventing Failed Extubations
Acronym: PreFIX
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00113877
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Ventilation Complication; Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extubated Patients: All patients receiving mechanical ventilation who are extubated in the intensive care units during the study period.
  Interventions: Diagnostic Test: Plateau Pressure

INTERVENTIONS:
Diagnostic Test: Plateau Pressure — Plateau pressure will be measured on all patients in the participating intensive care units prior to extubation.

SUMMARY:
More than 300,00 people in the United States experience acute respiratory failure and require mechanical ventilation every year. Of those that recover and are extubated, the most common reason for reintubation is recurrent respiratory failure. Our study proposes a novel methodology for identifying those patients most at risk for recurrent respiratory failure.

DETAILED DESCRIPTION:
Spontaneous breathing trials (SBTs) with pressure-support ventilation are commonly used to determine if mechanically ventilated patients are ready for extubation. However, 10-25% of all patients who pass a spontaneous breathing trial and are extubated will require re-intubation . Extubation failure is associated with an up to 50% increased risk of death independent of other risk factors and patient characteristics . Currently proposed methods for identifying patients who pass an SBT but are at high risk of reintubation perform poorly when applied in a real-world setting . Thus, there is a critical need to develop new methodologies for identifying patients at high risk for extubation failure.

Respiratory system mechanics, such as compliance, driving pressure, and plateau pressure, can identify patients at risk of poor outcomes, including prolonged mechanical ventilation and death. However, respiratory system mechanics are not commonly measured during spontaneous breathing trials, and the relationship between respiratory mechanics during an SBT and extubation failure is not known. This is due in part to long-standing concerns that accurate measurements of plateau pressures, and thus driving pressures and compliance, cannot be made in spontaneously breathing patients.

The objective of this study is to determine if respiratory compliance measured during a spontaneous breathing trial is a feasible method for identifying patients at increased risk of extubation failure.

ELIGIBILITY:
Inclusion Criteria:

* Extubated in participating ICU during study period

Exclusion Criteria:

* Previously extubated during hospitaliztion
* Extubation as part of transitioning to comfort measures

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All mechanically ventilated patients in participating intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who had a plateau pressure measured prior to extubation as a measure of feasibility | Day 0
  Feasibility is defined as 95% of patients having had a plateau pressure measured prior to extubation.

SECONDARY OUTCOMES:
Percentage of patients who were reintubated prior to hospital discharge | Day 0 to Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No